CLINICAL TRIAL: NCT02228915
Title: Analysis of Post-Translational Modifications of a Critical Protein Implicated in Amyotrophic Lateral Sclerosis
Acronym: SOD1
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1780
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2017-11

CONDITIONS: ALS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A portion of this sample will be stored for future use in study of ALS and how the critical protien affects the disease progression long term. This sample will be stored de-identified; therefore will not be linked to any identifying informaton about the subject. Sample will be stored at the UNC biophysics and Biochemistry lab indefinitely
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to discover and quantitate the differences in post-translational modifications found in the Cu, Zn superoxide dismutase (SOD1) of patients with amyotrophic lateral sclerosis (ALS) as compared to healthy individuals. SOD1 is a known genetic cause of ALS. With certain mutations, SOD1 gains a toxic function which leads to motor neuron death.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is a devastating neurodegenerative disease in which mutations in human Cu, Zn Superoxide Dismutase (SOD1) have been identified as a cause of familial ALS (FALS) cases.1-2 It has been shown that mutant SOD1 develops a novel toxic function through experiments demonstrating that many disease mutants maintain enzymatic activity, SOD1-null mice do not exhibit ALS symptoms, and co-expressed wild type protein does not rescue the disease-state.7-11 The majority of cases, however, are not caused directly by mutations of SOD1, instead being caused by a poorly understood interplay of several genes as well as environmental factors, which is often referred to as sporadic ALS (SALS).3 It has been found that FALS and SALS share similar pathology. 4-6 The hSOD1 protein aggregates characteristic of FALS have also been found in SALS patients, furthering the evidence that hSOD1 has an important role in the etiology of ALS in sporadic ALS patients.16-19 The exact mechanism of SOD1-associated toxicity has not yet been elucidated though many disease mutants have been shown to destabilize the SOD1 dimer. In this study we aim to compare the levels of SOD1 post-tra slational modifications in ALS patients to levels in healthy donors and to determine if there are distinct patterns of protein glutathionylation or phosphorylation. Our overall goal is to elucidate a direct mechanism of toxicity in SALS as well as identify potentially critical triggers

ELIGIBILITY:
Inclusion Criteria:

* SALS patients
* SOD1 associated FALS patients
* Healthy control

Exclusion Criteria: none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SALS patients SOD1 associated FALS patients Healthy control
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Post-translational modifications (PTMs) of Cu/Zn superoxide dismutase 1 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chafic Karam, MD, Principal Investigator — University of North Carolina, Chapel Hill; Nikolay V Dokholyan, PhD, Principal Investigator — UNC
Locations (1):
- UNC Neurology ALS clinic, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided